CLINICAL TRIAL: NCT07217652
Title: Investigating Mediodorsal Thalamus Representations Underlying Human Cognitive Flexibility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Hwang (Other)
Responsible Party: Sponsor-Investigator, Kai Hwang, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202412272
Record Dates: First submitted 2025-10-10; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: Cognitive control; working memory; decision making
MeSH Terms: conditions — Schizophrenia; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This is a within-subject research study. Each subject's performance on working memory, cognitive control, and decision-making functions will be compared across experimental conditions within each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within subject manipulation of working memory, cognitive control, and decision making (Experimental): Participants will complete a series of cognitive tasks designed to engage working memory, cognitive control, and decision-making. During these tasks, participants will view stimuli and make rule-based or value-based choices that require updating and applying context to guide behavior. Brain activity will be measured using high-resolution 7-Tesla functional MRI to assess how the mediodorsal thalamus and prefrontal cortex represent and update contextual information. Computational models will link behavior and neural activity to test how thalamic signals support flexible cognition and adaptive decision-making.
  Interventions: Other: High-resolution fMRI during working memory, cognitive control, and decision-making tasks

INTERVENTIONS:
Other: High-resolution fMRI during working memory, cognitive control, and decision-making tasks — Participants will perform a set of computerized cognitive tasks designed to test working memory, cognitive control, and decision-making while undergoing high-resolution 7-Tesla functional MRI. These tasks require participants to maintain and update contextual information, switch between rules, and make value-based choices under changing conditions. The intervention is distinguished by its integration of advanced neuroimaging with computational modeling to identify how the mediodorsal thalamus and prefrontal cortex represent, update, and generalize context. This approach allows precise mapping of thalamocortical mechanisms that support flexible cognition and goal-directed behavior.

SUMMARY:
The goal of this basic experimental research study is to examine how the human thalamus supports flexible thinking and behavior. Specifically, the research aims to elucidate how the mediodorsal (MD) thalamus encodes and updates "context"-the mental framework that determines which rules or actions are relevant in a given situation. This work may contribute to understanding why certain psychiatric conditions, such as schizophrenia and ADHD, involve difficulties with cognitive flexibility and control.

The primary research questions are:

Does the MD thalamus represent the context that organizes how working memory guides task selection? Does the MD thalamus signal when context needs to be updated after a change in task demands? Do these thalamic representations support generalization to new situations or rules?

Participants will complete cognitive tasks while undergoing high-resolution brain imaging using 7-Tesla MRI. The investigators will combine behavioral data, computational modeling, and advanced neuroimaging analyses to examine how the thalamus interacts with the cortex during flexible decision-making.

DETAILED DESCRIPTION:
The human brain's ability to learn and execute behaviors tailored to environmental contingencies is crucial for adaptive cognition. Central to this capacity are neural representations of context, which organize the associations between sensory features and behavioral utility. Despite their significance, the neural mechanisms underlying the encoding and updating of context representations remain poorly understood. This gap in knowledge is particularly relevant for understanding cognitive deficits in psychiatric disorders such as schizophrenia and ADHD.

This research study proposes to test the hypothesis that the human mediodorsal (MD) thalamus is critical for encoding, updating, and generalizing context representations. Previous studies have shown that damage to the MD thalamus impairs task switching and working memory in humans, consistent with findings from non-human animal models. Additionally, single-unit recordings in animals reveal that MD neurons rapidly encode task context, a process dependent on the convergence of prefrontal afferents. Preliminary fMRI data indicate that the human MD thalamus tracks task context and its updates following switches. However, a critical gap exists in interpreting these results due to the lack of quantitative models and advanced neuroimaging approaches to delineate the specific representations and computations carried out by the human MD.

To address this gap, the investigators will use a computational cognitive neuroscience approach, integrating computational models with high-resolution 7T MRI and advanced neuroimaging analyses. This study has three specific aims:

Aim 1: Determine whether the MD thalamus encodes context representations that organize how working memory guides task selection.

Aim 2: Investigate whether the MD thalamus encodes context prediction errors that flexibly switch prefrontal task representations.

Aim 3: Assess whether MD context representations enable generalization to novel stimulus-response contingencies during decision-making.

For all aims, the investigators will develop computational models that specify both cognitive processes and neural implementations to predict behavior and guide neuroimaging data analyses. This study aims to establish a new conceptual and empirical framework for understanding thalamic computation in humans, with significant implications for theories of cognitive control, adaptive human behavior, and cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* No history of any neurological, psychiatric, or medical condition that could affect cognition
* No use of benzodiazepines, long-acting opioids, or other psychotropic drugs that could alter cognitive performance
* Normal or corrected-to-normal vision (visual acuity)
* Normal color perception (Farnsworth-Munsell 100 Hue Test)
* Fluent in English
* No metal implants (including aneurysm clip, cardiac pacemaker, ICD, IUD, neurostimulation system, spinal cord stimulator, internal electrodes or wires, bone stimulator, ear implant, insulin or other infusion pump or device, prosthesis, artificial or prosthetic limb, shunt, vascular access port or catheter, thermodilution catheter, medication patch, radiation seeds or implants, wire mesh implant, tissue expander, surgical staples or clips or sutures, joint replacement, joint/bone pin/screw/nail/wire/plate, dentures, or non-removable hearing aid)
* No exposure to shrapnel or other-related MR contraindications
* No non-removable body piercing jewelry
* No non-removable makeup
* No history of claustrophobia
* No history of breathing problems
* Not currently pregnant or trying to get pregnant (this will be determined via self report and no records will be kept).

Exclusion Criteria:

* Has a history of any neurological, psychiatric, or medical condition that could affect cognition
* Use of benzodiazepines, long-acting opioids, or other psychotropic drugs that could alter cognitive performance
* Not fluent in English
* Known metal implants (including aneurysm clip, cardiac pacemaker, ICD, IUD, neurostimulation system, spinal cord stimulator, internal electrodes or wires, bone stimulator, ear implant, insulin or other infusion pump or device, prosthesis, artificial or prosthetic limb, shunt, vascular access port or catheter, thermodilution catheter, medication patch, radiation seeds or implants, wire mesh implant, tissue expander, surgical staples or clips or sutures, joint replacement, joint/bone pin/screw/nail/wire/plate, dentures, or non-removable hearing aid)
* History of claustrophobia
* Currently pregnant or trying to get pregnant (this will be determined via self report and no records will be kept).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Decoding of context representations in the medial dorsal thalamus from 7 T MRI data | Measured throughout the MRI session (approximately 90 minutes per participant).
  This outcome measure will quantify the extent to which multivariate patterns of brain activity in the MD thalamus encode task context. High-resolution 7-Tesla fMRI data will be analyzed using computational modeling and multivariate pattern analysis (MVPA) techniques.
  The primary metric will be decoding accuracy, expressed as a percentage ranging from 0% to 100%. Decoding accuracy reflects how well task contexts for working memory, cognitive control, and decision-making can be predicted from MD thalamic activity patterns. A value of 0% indicates chance-level or poor performance, while 100% indicates perfect prediction accuracy.
  For each participant, decoding accuracy will be computed as a single value using the same unit of measure (percentage accuracy). This value will reflect the overall ability to decode task context from MD activity and thus serves as the primary measure of this research study.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
This is a basic experimental study that involves human subjects; we do not publish our findings in ICMJE journals.

REFERENCES:
- [Background] Chen X, Leach SC, Hollis J, Cellier D, Hwang K. The thalamus encodes and updates context representations during hierarchical cognitive control. PLoS Biol. 2024 Dec 2;22(12):e3002937. doi: 10.1371/journal.pbio.3002937. eCollection 2024 Dec. PMID 39621781
- [Background] Shine JM, Lewis LD, Garrett DD, Hwang K. The impact of the human thalamus on brain-wide information processing. Nat Rev Neurosci. 2023 Jul;24(7):416-430. doi: 10.1038/s41583-023-00701-0. Epub 2023 May 26. PMID 37237103
- [Background] Hwang K, Bruss J, Tranel D, Boes AD. Network Localization of Executive Function Deficits in Patients with Focal Thalamic Lesions. J Cogn Neurosci. 2020 Dec;32(12):2303-2319. doi: 10.1162/jocn_a_01628. Epub 2020 Sep 9. PMID 32902335